CLINICAL TRIAL: NCT05085990
Title: A Phase 1a/b Dose Finding, Open-label Study to Evaluate Safety and Toxicity of Intravesical Instillation of TARA-002 in Adults with High-grade Non-muscle Invasive Bladder Cancer
Brief Title: Safety and Toxicity Study of Intravesical Instillation of TARA-002 in Adults with High-grade Non-muscle Invasive Bladder Cancer (Phase 1b)
Acronym: ADVANCED-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protara Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARA-002-101(Phase 1b)
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-09

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: Non-muscle invasive bladder cancer; bladder cancer; high grade Ta; carcinoma in situ; high-grade NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Intervention Model Description: All subjects will receive 6 weekly doses of TARA-002 at the recommended Phase 2 dose (R2PD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TARA-002 (Experimental): TARA-002 is a lyophilized biological preparation for instillation containing cells of Streptococcus pyogenes (Group A, type 3) Su strain treated with benzylpenicillin.
  Interventions: Biological: TARA-002

INTERVENTIONS:
Biological: TARA-002 — Phase 1b, Dose Expansion Phase: All subjects will receive 6 weekly doses of TARA-002 at the recommended Phase 2 dose (R2PD)

SUMMARY:
This study is open-label dose expansion study to investigate the safety and toxicity of intravesical treatment of high-grade NMIBC (HGTa or CIS, including CIS with concomitant Ta) after transurethral resection of bladder tumor (TURBT) and/or biopsy using TARA-002 in adults unable to obtain intravesical Bacillus Calmette-Guérin (BCG), adults who have received at least one dose of intravesical BCG or adults who have received at least one dose of intravesical chemotherapy.

After completion of the dose escalation phase (Phase 1a) and after the RP2D has been established, the dose expansion phase (Phase 1b) will start enrollment of subjects with CIS NMIBC with active disease to further evaluate the safety and preliminary efficacy of TARA-002, at the established RP2D. CIS NMIBC with active disease is defined as disease present at the last cystoscopic evaluation prior to signing the ICF. Subjects enrolled in the dose expansion phase will not include subjects previously enrolled and treated in the dose escalation phase.

All subjects will receive 6 weeks of treatment at the established RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older at the time of signing the informed consent
* Subjects who have voluntarily given written informed consent after the nature of the study has been explained according to applicable requirements prior to study entry
* Subjects with a histologically confirmed, high-grade Ta or CIS (including CIS with concomitant Ta) urothelial cell carcinoma of the bladder according to central review
* Subjects who are treatment naïve, unable to obtain intravesical BCG for the treatment of NMIBC, have received at least one dose of intravesical BCG, or at least one dose of intravesical chemotherapy

Exclusion Criteria:

* Penicillin allergy (subjects with a questionable history of allergy to penicillin or no history of penicillin use will undergo penicillin allergy testing prior to inclusion in the study)
* Predominant (defined as > 50%) adenocarcinoma, squamous cell carcinoma, or histological variants including plasmacytoid, sarcomatoid, or squamous components according to central review
* Concomitant prostatic or upper tract urothelial involvement per Investigator's assessment
* Nodal involvement or metastatic disease that existed at any time (past or present disease)
* Bladder cancer stage ≥ T1 within the last 36 months according to central histology review
* Bladder cancer stage CIS with concomitant T1

For more information on eligibility criteria, please contact the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Phase 1b, Dose Expansion Phase: Incidence of AEs in subjects with CIS NMIBC with active disease | Day 1 to Day 78
  AE = adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Operations Officer, Study Director — Protara Therapeutics
Locations (10):
- United States (10):
  - USC Norris Cancer Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Tulane Medical Center (TMC) - Clinic/Outpatient Facility, New Orleans, Louisiana
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - University of Rochester, Department of Urology, Rochester, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates PC, Nashville, Tennessee
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No